CLINICAL TRIAL: NCT01457534
Title: The Predictors for Continuous Renal Replacement Therapy in Liver Transplant Patient
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0671
Record Dates: First submitted 2011-10-04; First posted 2011-10-24 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver transplantation

SUMMARY:
Background. Acute renal failure after liver transplantation (LT) requiring continuous renal replacement therapy (CRRT) adversely affects patient survival. However, there are few reports to assess the predictors for postoperative CRRT in liver transplant patients. The investigators undertook this study to identify perioperative factors that would predict patients at risk of CRRT.

Patients and Methods. The investigators retrospectively reviewed the data of 148 liver transplant patients from January 2007 to November 2010 at Severance Hospital, Yonsei University HealthSystem, in Seoul, Korea. The number of patients treated with CRRT was 44 (18 patients from living and 26 from deceased donors) and those without CRRT was 104. Univariate and stepwise logistic multivariate analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65 year
* Liver transplant patients from January 2008 to December 2011

Exclusion Criteria:

* Patients treated with CRRT before transplantation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the data of 148 liver transplant patients from January 2008 to December 2011 at Severance Hospital, Yonsei University HealthSystem, in Seoul, Korea. The number of patients treated with CRRT was 44 (18 patients from living and 26 from deceased donors) and those without CRRT was 104.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
status before operation | 1 day before operation
  laboratory data(ex : total bilirubin, albumin, coagulation factors, blood gas analysis(arterial CO2 pressure. Blood urea nitrate/Creatinine, Hemoglobin/Hematocrit.)
the amount of ascites | intraoperative
the duration of anesthesia and operation | intraoperative
intraoperative hemodynamic instability | intraoperative
intraoperative bleeding | intraoperative
Intraoperative urine output | intraoperative
the types of donation(living or deceased donor) | intraoperative
survival rate | on the postoperative 28th days, 365 days
postoperative bleeding amount | on the postoperative 28th days, 365 days.
postoperative CRRT(continuous renal replacement therapy), | on the postoperative 28th days, 365days
mortality | on the postoperative 28th days, 365 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Wong LP, Blackley MP, Andreoni KA, Chin H, Falk RJ, Klemmer PJ. Survival of liver transplant candidates with acute renal failure receiving renal replacement therapy. Kidney Int. 2005 Jul;68(1):362-70. doi: 10.1111/j.1523-1755.2005.00408.x. PMID 15954928
- [Background] Wu CC, Yeung LK, Tsai WS, Tseng CF, Chu P, Huang TY, Lin YF, Lu KC. Incidence and factors predictive of acute renal failure in patients with advanced liver cirrhosis. Clin Nephrol. 2006 Jan;65(1):28-33. doi: 10.5414/cnp65028. PMID 16429839
- [Background] Gonwa TA, Mai ML, Melton LB, Hays SR, Goldstein RM, Levy MF, Klintmalm GB. Renal replacement therapy and orthotopic liver transplantation: the role of continuous veno-venous hemodialysis. Transplantation. 2001 May 27;71(10):1424-8. doi: 10.1097/00007890-200105270-00012. PMID 11391230
- [Background] Holt AW, Bierer P, Bersten AD, Bury LK, Vedig AE. Continuous renal replacement therapy in critically ill patients: monitoring circuit function. Anaesth Intensive Care. 1996 Aug;24(4):423-9. doi: 10.1177/0310057X9602400402. PMID 8862637
- [Background] Matsubara S, Okabe K, Ouchi K, Miyazaki Y, Yajima Y, Suzuki H, Otsuki M, Matsuno S. Continuous removal of middle molecules by hemofiltration in patients with acute liver failure. Crit Care Med. 1990 Dec;18(12):1331-8. doi: 10.1097/00003246-199012000-00005. PMID 2245605